CLINICAL TRIAL: NCT04409613
Title: Cost-Effectiveness Study on Establishing a Warfarin Counseling Clinic for Egyptian Patients With Mitral Valve Prostheses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Radwa Ahmed Batran, Doctor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ENREC-ASU.2019-99
Record Dates: First submitted 2020-05-24; First posted 2020-06-01 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Cost Effectiveness
MeSH Terms: interventions — Educational Status; Counseling

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical pharmacist-provided services+standard care group (Active Comparator): that receive clinical pharmacist-provided services at the Warfarin Counseling Clinic plus standard medical care
  Interventions: Other: Education and counseling
- Standard care group (No Intervention): that will receive standard medical care

INTERVENTIONS:
Other: Education and counseling — All patients or their caregivers will receive twenty minutes educational sessions for the first three visits according to patient ability to understand. At subsequent visits along the study duration, we will briefly review our educational material to refresh the patient's information. This will include: The objectives of treatment, disease progression process, risk factors, common symptoms of bleeding/thrombotic events and how to deal with this. Lifestyle modifications, including smoking cessation, blood pressure and diabetes control. Drug information: drug action, dose, indication, possible side effects, how to deal with the side effects, actions to take when missing the dose, storage conditions and when and how to administer. Possible interactions including drug-drug and drug-food interactions. Target INR and INR monitoring
  Arms: Clinical pharmacist-provided services+standard care group

SUMMARY:
The outcome of poor adherence to medications can be life threatening with certain drugs like warfarin. For each 10% increase in non-adherence to warfarin, there was a 14% increase in the risk of under-anticoagulation with significantly higher rates of morbidity and mortality. Furthermore, warfarin therapy is fraught with several inherent problems. These include a wide variation in dose requirement, delayed onset of anticoagulant effect, prolonged continuation after cessation of therapy, serious interactions with a wide range of medications and food items, risk of major hemorrhage related to overdosing, unpredictable control in presence of co-morbidities such as hepatic and renal impairment.

There is ongoing evidence that better outcomes are achieved when anticoagulation is managed by a pharmacist with expertise in anticoagulation management rather than usual care by physicians. Pharmacists can contribute to positive outcomes of therapy by educating and counseling patients to prepare and motivate them to follow their therapeutic regimens and monitoring plans, which will result substantially in improving the quality of care, reducing complications, and lowering hospitalization rates. Thus, beneficial effects of the pharmacist-managed counseling clinic have been repeatedly reported in terms of cost-effectiveness, patients' adherence to and knowledge about pharmacotherapy, and the outcome of treatment.

The objective of this study is to evaluate the cost-effectiveness of establishing a Medication Counseling Clinic for outpatients with mitral valve prostheses taking warfarin therapy in an Egyptian Teaching Hospital setting. Availability of this information could be used to target further quality improvement efforts, which may significantly improve outcomes for patients and cost containment efforts in an era when cost-effectiveness is at the forefront of healthcare policy initiatives.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (18-70) years.
2. Post mitral valve surgery patients.
3. Patients with a prescription of warfarin.

Exclusion Criteria:

1. Pregnant patients.
2. Patients with double and aortic valve replacement surgery.
3. Patients with biological prostheses.
4. Patients with congenital blood disorders.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Quality-adjusted life-years (QALYs) | 1 year
  The outcome of the two strategies will be measured in terms of quality-adjusted life-years (QALYs).This measurement weighs the length of life by the quality of life a patient experiences while in a specific health state. QALYs combine both morbidity and mortality into a single parameter.

CONTACTS AND LOCATIONS:
Overall Officials: Radwa Ahmed, Principal Investigator — Ain Shams University
Locations (1):
- Academy of CardioThoracic Surgery, Ain-Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Batran RA, Sabri NA, Ali I, Fahmy SF. Cost-Effectiveness of the Pharmacist-Managed Warfarin Therapy vs. Standard Care for Patients With Mechanical Mitral Valve Prostheses: An Egyptian Healthcare Perspective. Front Cardiovasc Med. 2022 Jul 13;9:889197. doi: 10.3389/fcvm.2022.889197. eCollection 2022. PMID 35911528